CLINICAL TRIAL: NCT02622750
Title: Triple-branch Stent Graft Placement and Total-arch Replacement for the Treatment of Acute DeBakey I Aortic Dissection: A Prospective, Multi-center, Randomized, Open-label, Parallel-group, Non-inferiority Clinical Trial
Brief Title: Triple-branch Stent Graft Placement and Total-arch Replacement for the Treatment of Acute DeBakey I Aortic Dissection
Acronym: TBSGPATART
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liang-Wan Chen MD (Other)
Collaborators: Xinqiao Hospital of Chongqing (Other); RenJi Hospital (Other); First Affiliated Hospital of Zhongshan Medical University (Other); Longyan City First Hospital (Other); The First City Hospital, ZhanZhou (Unknown)
Responsible Party: Sponsor-Investigator, Liang-Wan Chen MD, The director of the department of cardiovascular surgery, Fujian Medical University
Organization: Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLW2015AD2
Record Dates: First submitted 2015-11-19; First posted 2015-12-04 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2015-12

CONDITIONS: Acute Aortic Dissection
Keywords: triple-branched stent graft; total arch replace; the occluded rate of false lumen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- triple-branched stent graft (Experimental): The triple-branched stent graft was a branched 1-piece graft and included a main stent graft and 3 sidearm stent grafts (Yuhengjia Science and Technology, Corp, Ltd, Beijing, China). The main stent graft and sidearm stent grafts were individually mounted on 4 catheters and restrained by 4 silk sutures .The triple-branched stent graft was inserted into the true lumens of the aortic arch and proximal descending aorta; the three vascular stent branches were then grafted into the corresponding true lumens of the aortic arch branch vessels followed by the sequential release of the vascular stent backbone and the branch stents in the left subclavian artery, the left common carotid artery, and the innominate artery.
  Interventions: Procedure: triple-branched stent graft
- four-branched Dacron graft (Active Comparator): A four-branched Dacron graft (Boston Scientific Inc, Boston, MA) and a stent graft (MicroPort Medical Co Ltd, Shanghai, China) were used in total arch replacement combined with stented elephant trunk (SET) implantation.The SET was inserted into the true lumen of the descending aorta.The proximal edge of the residual aorta was trimmed to match the proximal end of the stent graft.The anastomosis between the four-branched prosthetic graft and the distal aorta containing the intraluminal stented graft was carried out using "open" aortic technique.
  Interventions: Procedure: four-branched Dacron graft

INTERVENTIONS:
Procedure: triple-branched stent graft — place the triple-branched stent graft into the aortic arch, descending aorta ,the left subclavian artery, the left common carotid artery, and the innominate artery.
  Arms: triple-branched stent graft
Procedure: four-branched Dacron graft — The stent elephant trunk was inserted into the true lumen of the distal aorta in a bound, compressed state after the distal aorta was transected between the origin of the left subclavian artery and the left carotid artery. The distal aorta incorporating the stent graft was firmly attached to the distal end of the four-branched Dacron graft using the "open" aortic procedure. After the anastomosis was completed, blood perfusion of the lower body was started via the perfusion limb of the four-branched Dacron graft.
  Arms: four-branched Dacron graft

SUMMARY:
The purpose of this study is to compare triple-branched stent placement with total-arch replacement in the treatment of acute DeBakey I aortic dissection . The investigators design optimal effect compare prospective, multi-center, randomized, open-label, parallel-group, non-inferiority clinical trial.

DETAILED DESCRIPTION:
From November 2015, 90 consecutive patients with acute DeBakey I aortic dissection from five-centers in China were treated with triple-branched stent placement or hemi-arch replacement. The distribution of the patients adopts the dynamic random variance minimization random method. About half of the patients will be assigned to the the stent-graft group, the other to the hemi-arch group.

In all cases, surgery was performed under general anesthesia with tracheal intubation and cardiopulmonary bypass (CPB). During surgery arterial pressures at the upper and lower limbs were monitored. An esophageal echocardiography probe was placed routinely, and a sternal incision was performed. To establish CPB, the perfusion tube was placed in the right axillary artery and the drainage tube was placed in the superior and inferior vena cava through the right atrium. The CPB flow rate was of 2.4-2.6 L/kg/min. Intermittent cold blood cardioplegia was perfused through the left and right coronary arteries for myocardial protection.

In stent-graft group , the innominate artery and the left common carotid artery were fully isolated during the CPB cooling process. The ascending aorta proximal to the innominate artery was occluded, and the ascending aorta was transected slightly above the sinus tube connection; the left and right coronary arteries were directly perfused with blood-containing cold cardioplegia. Proximal procedures such as aortic valve repair, sinus reconstruction, and root replacement were performed first. Afterwards, the stumps were reconstructed. The reconstructed aortic root stump was anastomosed with a Dacron graft of corresponding size using 4-0 polypropylene suture (ascending aorta replacement). The nasopharyngeal temperature was then decreased to 25° (usually a rectal temperature of 27-29°C), the aortic perfusion flow was set to 10-15 ml/kg/min, and the innominate artery and the left common carotid artery were occluded 5-6 cm above the aortic arch. The aortic occlusion clamp was removed and a half aortic arch transection was made about 2 cm proximal to the innominate artery. Through the incision, the true lumens of the aortic arch, the proximal descending aorta, and the three aortic branches were identified. The triple-branched stent graft was inserted into the true lumens of the aortic arch and proximal descending aorta; the three stent graft branches were then placed into the corresponding true lumens of the aortic arch branch vessels followed by the sequential release of the vascular stent backbone and the branch stents in the left subclavian artery, the left common carotid artery, and the innominate artery. A catheter with a balloon or a probe was used to expand the vascular stents and the graft and branches were examined for kinks or folding of the backbone. A sandwich reconstruction was performed between the aortic stump, the aortic external Dacron graft, and the proximal stentless suture zone of the intraluminal artificial vessel backbone. The reconstructed stump was anastomosed with the Dacron graft that replaced the ascending aorta using 4-0 polypropylene suture. The occlusions of the left common carotid artery and the innominate artery were then relieved, and air was fully flushed out from the heart and the aorta. The right axillary artery perfusion was stopped, and systemic perfusion via an aortic perfusion tube at the artificial portion of the ascending aorta was performed. The patient was rewarmed after oxygen debt repayment, followed by the cardiac resuscitation.

In total-arch group , the ascending aorta proximal to the innominate artery was blocked during the CPB cooling process, and the ascending aorta was incised and transected slightly above the sinus tube connection. The left and right coronary arteries were directly perfused with blood-containing cold cardioplegia. As in stent-graft group , proximal procedures were performed first. The reconstructed aortic root stumps were sutured with Dacron graft using 4-0 polypropylene suture (ascending aorta replacement). The nasopharyngeal temperature was then decreased to 25° (usually a rectal temperature of 27-29°C) and the aortic perfusion flow was set to 10-15 ml/kg/min. The innominate artery and the left common carotid artery were clamped 5-6 cm above the aortic arch and the aortic occlusion clamp was removed. Half aortic arch resection was performed along the greater curvature of the aortic arch at 1 cm proximal of the innominate artery to the lesser curvature of the aortic arch at the origin of the descending aorta. Stumps between the dissection slices were lined with cotta slices and reconstructed using the sandwich method and then anastomosed with an Dacron graft of the corresponding size and shape using 4-0 polypropylene suture. Finally, the proximal end was anastomosed with the artificial blood vessel using 4-0 polypropylene suture. Air was fully flushed from the heart and aorta. The right auxiliary artery perfusion was stopped and systemic perfusion via an aortic perfusion tube at the artificial blood vessel of the ascending aorta was performed. The patient was rewarmed after oxygen debt repayment, followed by cardiac resuscitation.

Telephone contact was maintained with the patients after discharge. At 3,6,12 months postoperatively , patients received a follow-up examination, chest radiography, echocardiography, bilateral carotid artery Doppler examinations and CT angiography (CTA) examinations Numerical data were expressed as percentages, and comparisons between groups were performed with the chi-square test. Quantitative data were expressed as mean ± standard deviation; the independent sample t test was used for group comparisons and the paired t-test was used to compare the groups before and after surgery. The primary end point is the occluded rate of the false lumen one year postoperatively. The secondary end point are the survive rate ,complication, reoperation rate, the growth rate of thoracic descending aorta, security index perioperatively, life quality postoperatively.Statistical analysis were performed with SPSS 11.5 software. A value of P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age<65 years
* acute DeBakkey I aortic dissection is confirmed by CTA
* cardiac function is NYHA I-II
* the onset time< 2 weeks
* the patient or family members can understand the research plan and will participate in this study and provide a written informed consent

Exclusion Criteria:

* Dissection involved the superior mesenteric artery, renal artery and coronary artery, which affect the body's viscera function seriously. The principal researcher from different centre need judge the patients' condition.
* there is a serious complication of nervous system, such as coma, paraplegia, etc
* pregnant or lactating women
* anyone with severe emphysema, interstitial pneumonia or ischemic heart disease cannot tolerate surgery
* subjects with contraindications of heart surgery, anesthesia and extracorporeal circulation
* subjects had significant or progressive of heart disease, according to the experience of the researchers,whose life expectancy is less than 1 year, or placement of triple- branched stent graft will induce unacceptable risk to the subjects
* anyone with serious mental illness, drug abuse, alcoholism, prison inmates, a lack of ability to care for, or can not express the informed consent
* subjects are incompliance or can't complete the research
* anyone is involved in the other clinical trial
* other reasons are not suitable for clinical trials, according to the researchers

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
the occluded rate of false lumen by the CTA | 1 year postoperatively

SECONDARY OUTCOMES:
the survive rate by the questionnaire | 3 months, 6 months, 12 months postoperatively
complication by the datum of case | 1 months postoperatively
reoperation rate by the datum of case | 1 year postoperatively
the growth rate of thoracic descending aorta by the CTA | 3 months, 6 months, 12 months postoperatively
security index by the datum of case | 7 days perioperatively
life quality by the questionnaire | 3 months, 6 months, 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Wan Chen, M.D PH, Study Director — the director of the department of cardiovascular surgery Union Hospital FuJian Medical University
Locations (1):
- the Department of Cardiovascular Surgery, Fuzhou, Fujian, China

REFERENCES:
- [Background] Chen LW, Dai XF, Lu L, Zhang GC, Cao H. Extensive primary repair of the thoracic aorta in acute type a aortic dissection by means of ascending aorta replacement combined with open placement of triple-branched stent graft: early results. Circulation. 2010 Oct 5;122(14):1373-8. doi: 10.1161/CIRCULATIONAHA.110.946012. Epub 2010 Sep 20. PMID 20855660
- [Background] Chen LW, Wu XJ, Lu L, Zhang GC, Yang GF, Yang ZW, Dong Y, Cao H, Chen Q. Total arch repair for acute type A aortic dissection with 2 modified techniques: open single-branched stent graft placement and reinforcement of the dissected arch vessel stump with stent graft. Circulation. 2011 Jun 7;123(22):2536-41. doi: 10.1161/CIRCULATIONAHA.110.008656. Epub 2011 May 16. PMID 21576657
- [Background] Sun L, Qi R, Chang Q, Zhu J, Liu Y, Yu C, Zhang H, Lv B, Zheng J, Tian L, Lu J. Surgery for marfan patients with acute type a dissection using a stented elephant trunk procedure. Ann Thorac Surg. 2008 Dec;86(6):1821-5. doi: 10.1016/j.athoracsur.2008.08.026. PMID 19021985
- [Background] Sun L, Qi R, Chang Q, Zhu J, Liu Y, Yu C, Zhang H, Lv B, Zheng J, Tian L, Lu J. Surgery for acute type A dissection with the tear in the descending aorta using a stented elephant trunk procedure. Ann Thorac Surg. 2009 Apr;87(4):1177-80. doi: 10.1016/j.athoracsur.2009.01.042. PMID 19324146
- [Background] Liu ZG, Sun LZ, Chang Q, Zhu JM, Dong C, Yu CT, Liu YM, Zhang HT. Should the "elephant trunk" be skeletonized? Total arch replacement combined with stented elephant trunk implantation for Stanford type A aortic dissection. J Thorac Cardiovasc Surg. 2006 Jan;131(1):107-13. doi: 10.1016/j.jtcvs.2005.09.015. Epub 2005 Dec 9. PMID 16399301
- [Background] Estrera AL, Miller CC 3rd, Huynh TT, Porat E, Safi HJ. Neurologic outcome after thoracic and thoracoabdominal aortic aneurysm repair. Ann Thorac Surg. 2001 Oct;72(4):1225-30; discussion 1230-1. doi: 10.1016/s0003-4975(01)02971-x. PMID 11603441
- [Background] Chiappini B, Schepens M, Tan E, Dell' Amore A, Morshuis W, Dossche K, Bergonzini M, Camurri N, Reggiani LB, Marinelli G, Di Bartolomeo R. Early and late outcomes of acute type A aortic dissection: analysis of risk factors in 487 consecutive patients. Eur Heart J. 2005 Jan;26(2):180-6. doi: 10.1093/eurheartj/ehi024. Epub 2004 Dec 7. PMID 15618075
- [Background] Trimarchi S, Nienaber CA, Rampoldi V, Myrmel T, Suzuki T, Mehta RH, Bossone E, Cooper JV, Smith DE, Menicanti L, Frigiola A, Oh JK, Deeb MG, Isselbacher EM, Eagle KA; International Registry of Acute Aortic Dissection Investigators. Contemporary results of surgery in acute type A aortic dissection: The International Registry of Acute Aortic Dissection experience. J Thorac Cardiovasc Surg. 2005 Jan;129(1):112-22. doi: 10.1016/j.jtcvs.2004.09.005. PMID 15632832
- [Background] Rampoldi V, Trimarchi S, Eagle KA, Nienaber CA, Oh JK, Bossone E, Myrmel T, Sangiorgi GM, De Vincentiis C, Cooper JV, Fang J, Smith D, Tsai T, Raghupathy A, Fattori R, Sechtem U, Deeb MG, Sundt TM 3rd, Isselbacher EM; International Registry of Acute Aortic Dissection (IRAD) Investigators. Simple risk models to predict surgical mortality in acute type A aortic dissection: the International Registry of Acute Aortic Dissection score. Ann Thorac Surg. 2007 Jan;83(1):55-61. doi: 10.1016/j.athoracsur.2006.08.007. PMID 17184630
- [Background] Crawford ES, Kirklin JW, Naftel DC, Svensson LG, Coselli JS, Safi HJ. Surgery for acute dissection of ascending aorta. Should the arch be included? J Thorac Cardiovasc Surg. 1992 Jul;104(1):46-59. PMID 1614214
- [Background] Hirotani T, Nakamichi T, Munakata M, Takeuchi S. Routine extended graft replacement for an acute type A aortic dissection and the patency of the residual false channel. Ann Thorac Surg. 2003 Dec;76(6):1957-61. doi: 10.1016/s0003-4975(03)01325-0. PMID 14667621
- [Background] Takahara Y, Sudo Y, Mogi K, Nakayama M, Sakurai M. Total aortic arch grafting for acute type A dissection: analysis of residual false lumen. Ann Thorac Surg. 2002 Feb;73(2):450-4. doi: 10.1016/s0003-4975(01)03422-1. PMID 11845858
- [Background] Urbanski PP, Siebel A, Zacher M, Hacker RW. Is extended aortic replacement in acute type A dissection justifiable? Ann Thorac Surg. 2003 Feb;75(2):525-9. doi: 10.1016/s0003-4975(02)04378-3. PMID 12607666
- [Background] Khan IA, Nair CK. Clinical, diagnostic, and management perspectives of aortic dissection. Chest. 2002 Jul;122(1):311-28. doi: 10.1378/chest.122.1.311. PMID 12114376
- [Background] Pochettino A, Brinkman WT, Moeller P, Szeto WY, Moser W, Cornelius K, Bowen FW, Woo YJ, Bavaria JE. Antegrade thoracic stent grafting during repair of acute DeBakey I dissection prevents development of thoracoabdominal aortic aneurysms. Ann Thorac Surg. 2009 Aug;88(2):482-9; discussion 489-90. doi: 10.1016/j.athoracsur.2009.04.046. PMID 19632398
- [Background] Zierer A, Voeller RK, Hill KE, Kouchoukos NT, Damiano RJ Jr, Moon MR. Aortic enlargement and late reoperation after repair of acute type A aortic dissection. Ann Thorac Surg. 2007 Aug;84(2):479-86; discussion 486-7. doi: 10.1016/j.athoracsur.2007.03.084. PMID 17643619
- [Background] Halstead JC, Meier M, Etz C, Spielvogel D, Bodian C, Wurm M, Shahani R, Griepp RB. The fate of the distal aorta after repair of acute type A aortic dissection. J Thorac Cardiovasc Surg. 2007 Jan;133(1):127-35. doi: 10.1016/j.jtcvs.2006.07.043. Epub 2006 Dec 4. PMID 17198797
- [Background] Park KH, Lim C, Choi JH, Chung E, Choi SI, Chun EJ, Sung K. Midterm change of descending aortic false lumen after repair of acute type I dissection. Ann Thorac Surg. 2009 Jan;87(1):103-8. doi: 10.1016/j.athoracsur.2008.09.032. PMID 19101279
- [Background] Jakob H, Tsagakis K, Tossios P, Massoudy P, Thielmann M, Buck T, Eggebrecht H, Kamler M. Combining classic surgery with descending stent grafting for acute DeBakey type I dissection. Ann Thorac Surg. 2008 Jul;86(1):95-101. doi: 10.1016/j.athoracsur.2008.03.037. PMID 18573404
- [Background] Uchida N, Shibamura H, Katayama A, Shimada N, Sutoh M, Ishihara H. Operative strategy for acute type a aortic dissection: ascending aortic or hemiarch versus total arch replacement with frozen elephant trunk. Ann Thorac Surg. 2009 Mar;87(3):773-7. doi: 10.1016/j.athoracsur.2008.11.061. PMID 19231387
- [Background] Gorlitzer M, Weiss G, Meinhart J, Waldenberger F, Thalmann M, Folkmann S, Moidl R, Grabenwoeger M. Fate of the false lumen after combined surgical and endovascular repair treating Stanford type A aortic dissections. Ann Thorac Surg. 2010 Mar;89(3):794-9. doi: 10.1016/j.athoracsur.2009.11.054. PMID 20172130
- [Background] Mizuno T, Toyama M, Tabuchi N, Wu H, Sunamori M. Stented elephant trunk procedure combined with ascending aorta and arch replacement for acute type A aortic dissection. Eur J Cardiothorac Surg. 2002 Oct;22(4):504-9. doi: 10.1016/s1010-7940(02)00429-3. PMID 12297163
- [Background] Kazui T, Washiyama N, Muhammad BA, Terada H, Yamashita K, Takinami M, Tamiya Y. Total arch replacement using aortic arch branched grafts with the aid of antegrade selective cerebral perfusion. Ann Thorac Surg. 2000 Jul;70(1):3-8; discussion 8-9. doi: 10.1016/s0003-4975(00)01535-6. PMID 10921673
- [Background] Czerny M, Zimpfer D, Fleck T, Hofmann W, Schoder M, Cejna M, Stampfl P, Lammer J, Wolner E, Grabenwoger M. Initial results after combined repair of aortic arch aneurysms by sequential transposition of the supra-aortic branches and consecutive endovascular stent-graft placement. Ann Thorac Surg. 2004 Oct;78(4):1256-60. doi: 10.1016/j.athoracsur.2004.03.063. PMID 15464481